CLINICAL TRIAL: NCT06089408
Title: Weighted Blanket Use in Oncology Patients to Reduce Anxiety
Brief Title: Weighted Blanket Use to Reduce Anxiety in Oncology Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Allison De Villiers, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-22313; NCI-2023-06974 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-09-27; First posted 2023-10-18 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (weighted blanket) (Experimental): Patients use a weighted blanket for 30 minutes during the infusion appointment.
  Interventions: Other: Supportive Care; Other: Survey Administration
- Arm II (regular blanket) (Active Comparator): Patients use a regular blanket for 30 minutes per standard of care during the infusion appointment.
  Interventions: Other: Best Practice; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Use a regular blanket
  Other Names: standard of care; standard therapy
  Arms: Arm II (regular blanket)
Other: Supportive Care — Use a weighted blanket
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: Arm I (weighted blanket)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial compares the effect of using weighted blankets versus regular blankets during first time infusions (e.g. chemotherapy, targeted therapy etc.) to decrease adverse side effects such as anxiety and distress in cancer (oncology) patients. Feeling safe, comforted, and grounded in the world are some of the benefits noted by individuals who use weighted blankets. Deep touch pressure (DTP) has been found to reduce symptoms of stress and anxiety and is defined as a sensation one feels when being hugged, squeezed, or held. DTP affects the nervous system by creating a calming effect which may lower stress and increase feelings of well-being. The use of weighted blankets may help to manage anxiety and distress during chemotherapy or immunotherapy infusions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the efficacy of weighted blankets on anxiety in patients receiving infusion therapy.

SECONDARY OBJECTIVE:

I. To assess the efficacy of weighted blankets on distress in patients receiving infusion therapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients use a weighted blanket for 30 minutes during the infusion appointment.

ARM II: Patients use a regular blanket for 30 minutes per standard of care during the infusion appointment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age and older
* About to begin either targeted or cytotoxic chemotherapy
* Able to comprehend and sign a consent form
* Able to read and complete surveys
* Alert and oriented

Exclusion Criteria:

* Currently using a weighted blanket at home
* Non-English speaking
* Peripheral neuropathy
* Fibromyalgia
* Open pressure ulcer
* Recent surgical flap
* Claustrophobic
* Weight 45 kg or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Levels of anxiety using State Trait Anxiety Inventory (STAI) for Adults, short form | At baseline and 30 minutes after use of either a standard or weighted blanket
  To test for the effect of the weighted blanket, will fit a mixed model with the post-level of anxiety as the dependent variable and baseline values and treatment (standard or weighted blanket) as predictors. A random effect for patient will be fit to account for the possible correlation of within-patient repeated outcome measures. The models will control for patient gender and age.

SECONDARY OUTCOMES:
Levels of distress using NCCN Distress Thermometer | At baseline and 30 minutes after use of either a standard or weighted blanket
  To test for the effect of the weighted blanket, will fit a mixed model with the post-level of distress as the dependent variable and baseline values and treatment (standard or weighted blanket) as predictors. A random effect for patient will be fit to account for the possible correlation of within-patient repeated outcome measures. The models will control for patient gender and age.
Qualitative change in levels of anxiety based on the baseline and 30 min post blanket use scores using State Trait Anxiety Inventory (STAI) for Adults, short form | At baseline and 30 minutes after use of either a standard or weighted blanket
  Will be binned to create ordinal variables. If they lead to an adequate sample size in each group, clinically relevant cut points will be used for binning. Otherwise, we will bin using outcome medians or terciles, with the choice depending on the distribution of the data collected after blanket use. The categorical representation will be modeled using generalized linear mixed modeling. We will fit ordinal logistic regression models with repeated measures. As with the linear mixed models, baseline values and treatment (standard or weighted blanket) will be predictors, with patient gender and age as control variables.
Qualitative change in levels of distress based on the baseline and 30 min post blanket use scores using NCCN Distress Thermometer | At baseline and 30 minutes after use of either a standard or weighted blanket
  Will be binned to create ordinal variables. If they lead to an adequate sample size in each group, clinically relevant cut points will be used for binning. Otherwise, we will bin using outcome medians or terciles, with the choice depending on the distribution of the data collected after blanket use. The categorical representation will be modeled using generalized linear mixed modeling. We will fit ordinal logistic regression models with repeated measures. As with the linear mixed models, baseline values and treatment (standard or weighted blanket) will be predictors, with patient gender and age as control variables.

CONTACTS AND LOCATIONS:
Overall Officials: Allison De Villiers, MSN, RN, ONC, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu